CLINICAL TRIAL: NCT00027703
Title: A Double Blind, Placebo Controlled Randomized Phase II Trial Of Gemcitabine And Cisplatin With Or Without The VEGF Inhibitor Bevacizumab (NSC #704865) In Patients With Malignant Mesotheloma
Brief Title: Combination Chemotherapy With or Without Bevacizumab in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02430; NCI-2012-02430 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069058; NCI-2710; UCCRC-11046A; 11046A (Other: University of Chicago); 2710 (Other: CTEP); N01CM17102 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2012-12

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Localized Malignant Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Gemcitabine; Cisplatin; Bevacizumab

ARMS (2):
- Arm I (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 30-60 minutes (beginning after gemcitabine infusion) and bevacizumab IV over 30-90 minutes (beginning after cisplatin infusion) on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease (SD), complete response (CR), or partial response (PR) after the sixth course may receive bevacizumab as a single agent once every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: cisplatin; Biological: bevacizumab; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive gemcitabine and cisplatin as in arm I and placebo IV over 30-90 minutes (beginning after cisplatin infusion) on day 1. Treatment repeats as in arm I. Patients who achieve SD, CR, or PR after the sixth course may receive placebo as a single agent once every 3 weeks in the absence of disease progression.
  Interventions: Drug: gemcitabine hydrochloride; Drug: cisplatin; Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm I
Other: placebo — Given IV
  Other Names: PLCB
  Arms: Arm II
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is to see if combination chemotherapy works better with or without bevacizumab in treating patients who have malignant mesothelioma. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. It is not yet known if combination chemotherapy works better with or without bevacizumab in treating malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the time to progression of patients with malignant mesothelioma treated with gemcitabine and cisplatin with or without bevacizumab.

II. Compare the objective response rate in patients treated with these regimens.

III. Compare the toxicity of these regimens when administered to these patients.

IV. Compare the median and overall survival of patients treated with these regimens.

V. Assess plasma vascular endothelial growth factor and serum vascular cell adhesion molecule-1 levels before, during, and after study therapy as predictors of outcome in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to histology (epithelial vs other) and ECOG performance status (0 vs 1). Patients are randomized to one of two treatment arms.

ARM I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 30-60 minutes (beginning after gemcitabine infusion) and bevacizumab IV over 30-90 minutes (beginning after cisplatin infusion) on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease (SD), complete response (CR), or partial response (PR) after the sixth course may receive bevacizumab as a single agent once every 3 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive gemcitabine and cisplatin as in arm I and placebo IV over 30-90 minutes (beginning after cisplatin infusion) on day 1. Treatment repeats as in arm I. Patients who achieve SD, CR, or PR after the sixth course may receive placebo as a single agent once every 3 weeks in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant pleural or peritoneal mesothelioma that is not amenable to curative surgery

  * Epithelial, sarcomatoid, or mixed subtype
  * Evidence of gross unresectability, including, but not limited to, the following conditions:

    * Direct extension into the chest wall
    * Mediastinal or hilar lymphadenopathy
    * Pulmonary or cardiac function that is inadequate to tolerate resection
    * Sarcomatoid or mixed histology
* Pleural mesothelioma must be stage II or greater using the International Mesothelioma Interest Group staging system
* Measurable disease outside prior irradiation port

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Pleural effusions and ascites are not considered measurable lesions
  * Site in pleura, lung, liver, or retroperitoneum that can be assessed by MRI for evaluation of blood flow
* No obvious tumor involvement of major vessels by CT scan
* No known brain metastases
* Performance status - ECOG 0-1
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of bleeding diathesis
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* INR no greater than 1.5
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* If 1+ or greater proteinuria on dipstick, then must have less than 500 mg of protein/24-hour urine collection
* No significant renal impairment
* See Disease Characteristics
* No history deep vein thrombosis
* No myocardial ischemia or infarction within the past 6 months
* No uncompensated coronary artery disease within the past 6 months
* No uncontrolled hypertension
* No symptomatic congestive heart failure
* No unstable angina pectoris within the past 6 months
* No cardiac arrhythmia
* No transient ischemic attack within the past 6 months
* No cerebrovascular accident within the past 6 months
* No other arterial thromboembolic event within the past 6 months
* No clinically significant peripheral artery disease
* See Disease Characteristics
* No history of pulmonary embolism
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or other study agents
* No other active malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No ongoing or active infection
* No other concurrent uncontrolled illness that would preclude study participation
* No psychiatric illness or social situations that would preclude compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No growth factors for 24 hours before, during, or for 24 hours after cytotoxic chemotherapy
* See Biologic therapy
* Prior intrapleural cytotoxic agents (including bleomycin) allowed
* No prior systemic cytotoxic chemotherapy
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* See Disease Characteristics
* At least 6 weeks since prior major surgery
* At least 30 days since prior investigational drug
* No other concurrent investigational or commercial agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2001-10; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | Time from randomization until the first evidence of progression, up to 9 years
  The two treatment groups will be compared using a stratified logrank test. Kaplan-Meier time-to-event curves will be constructed for each treatment group. Median time-to-progression in each group and corresponding 95% confidence intervals will be derived using the method described in Brookmeyer and Crowley.

SECONDARY OUTCOMES:
Complete response rate | Up to 6 months
  Will be compared between groups using chi-square or Fisher exact tests, as appropriate.
Objective response rate (complete and partial response) | Up to 6 months
  Will be compared between groups using chi-square or Fisher exact tests, as appropriate.
Rate of disease stabilization | Up to 6 months
  Will be compared between groups using chi-square or Fisher exact tests, as appropriate.
Overall survival | Up to 9 years
  Kaplan-Meier estimates of overall survival rates will be derived and compared between the two groups using a stratified log-rank test.
Incidence of adverse events graded according to NCI CTCAE version 3.0 | Up to 9 years
  Toxicity rates will be compared between the two groups via chi-square or Fisher exact tests.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States